CLINICAL TRIAL: NCT00985933
Title: A Single Center, Double-Blind, Randomized, Double Dummy, Placebo-Controlled, Three-Period Crossover Study to Assess the Effects of a mGluR2/3 Positive Allosteric Modulator [AZD8529] Upon Ketamine-Induced Cortical Stimulation and Impairment of Working-Memory Related Activation of the Prefrontal Cortex
Brief Title: The Effects AZD8529 on Ketamine-induced Impairment of Working Memory in Healthy Volunteers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D2285M00015
Record Dates: First submitted 2009-09-25; First posted 2009-09-29 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-05

CONDITIONS: Healthy; Memory Impairment
Keywords: Healthy normal volunteers
MeSH Terms: conditions — Memory Disorders | interventions — AZD8529

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental): 180 mg of AZD8529
  Interventions: Drug: AZD8529; Drug: Placebo to match AZD8529
- 2 (Experimental): 50 mg AD8529
  Interventions: Drug: AZD8529; Drug: Placebo to match AZD8529
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: AZD8529; Drug: Placebo to match AZD8529

INTERVENTIONS:
Drug: AZD8529 — 6 capsules by mouth 1 time 12 to 24 prior to assessments
Drug: Placebo to match AZD8529 — 6 capsules by mouth 1 time 12 to 24 hours prior to assessments

SUMMARY:
The purpose of this study is to assess if ketamine will induce, in healthy volunteers, impairment of working memory and if the drug AZD8529 will block the effects of ketamine on working memory as assessed by functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

* Right handed
* 12th grade education or equivalent
* Able to read and write English as primary language

Exclusion Criteria:

* History of head injury
* Substance abuse or dependence
* History of claustrophobia

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
fMRI | 3
Ketamine Infusion | 3

SECONDARY OUTCOMES:
Clinician Administered Dissociative States Scale (CADSS)
Positive and Negative Syndrome Scale (PANSS)
Laboratory assessment: electrocardiogram (ECG), physical exam, vital signs, collection of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: John Krystal, Principal Investigator — Chair, Department of PsychiatryYale University School of MedicineChief of Psychiatry, Yale-New Haven Hospital
Locations (1):
- Research Site, New Haven, Connecticut, United States